CLINICAL TRIAL: NCT00189904
Title: A Multicenter, Open-label Phase I/II Study to Evaluate Safety and Immunogenicity of MVA-BN® Smallpox Vaccine in HIV Infected Subjects (CD4 Counts >350 / µl) and Healthy Subjects With and Without Previous Smallpox Vaccination
Brief Title: Safety, Tolerability and Immune Response of IMVAMUNE (MVA-BN)Smallpox Vaccine in HIV Infected Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: POX-MVA-010; HHSN266200400072C
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2007-12

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

INTERVENTIONS:
Biological: IMVAMUNE (MVA-BN)

SUMMARY:
The purpose of this study is to gather information on the safety and immunogenicity of an investigational smallpox vaccine in HIV infected populations.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between 18 and 49 years of age or female subjects between 18 and 55 years of age who provided informed consent.
* Women with negative pregnancy test.
* Women of childbearing potential must use an acceptable method of contraception.
* Cardiac enzymes within ULN.
* White blood cells ≥ 2500/mm3 and < 11,000/ mm3.
* Absolute neutrophil count ≥ 1000/mm3.
* Adequate renal function.
* Adequate hepatic function.
* Negative hepatitis B surface antigen (HBsAg) and hepatitis B core antibody (anti-HBc).
* Negative antibody test to hepatitis C virus (HCV).
* Negative urine glucose by dipstick or urinalysis.
* Normal 12-lead electrocardiogram.
* Availability for follow-up during the study.

Groups 1 and 3 (All vaccinia-naïve subjects) additionally:

* No history of known or suspected previous smallpox vaccination.
* No detectable vaccinia scar.
* No military service prior to 1989 or after January 2003.

Groups 2 and 4 (All previously vaccinated subjects) additionally:

* History of at least one previous smallpox vaccination
* Time since most current smallpox vaccination > 10 years.

Groups 1 and 2 (All HIV Infected subjects) additionally:

* Documented HIV-1 infection
* Plasma HIV-1 RNA level < 400 copies/mL at screening.
* CD4 cells ≥ 350/µL
* Haemoglobin ≥ 9.0 g/dL.
* Platelets ≥ 100,000/mm3.
* AST (SGOT), ALT (SGPT) and alkaline phosphatase ≤ 3 x ULN

Groups 3 and 4 (All Healthy subjects) additionally:

* Negative ELISA for HIV.
* Haemoglobin >11 g/dL.
* Platelets ≥ 140,000/mm3.
* AST (SGOT), ALT (SGPT) and alkaline phosphatase without clinically significant findings

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Uncontrolled serious infection i.e. not responding to antimicrobial therapy.
* History of any serious medical condition (other than HIV infection).
* History of or active autoimmune disease.
* Known or suspected impairment of immunologic function (other than HIV infection).
* History of malignancy.
* History or clinical manifestation of clinically significant and severe haematological, renal, hepatic, pulmonary, central nervous, cardiovascular or gastrointestinal disorders.
* Clinically significant mental disorder not adequately controlled by medical treatment.
* Any condition which might interfere with study objectives.
* History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, or any other heart condition under the care of a doctor.
* History of an immediate family member with onset of ischemic heart disease before age 50.
* Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool.
* History of chronic alcohol abuse and/or intravenous drug abuse.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Known previous allergic reaction to immunoglobulins.
* Known allergies to cidofovir or probenecid.
* History of anaphylaxis or severe allergic reaction.
* Acute disease (illness with or without a fever) at the time of enrollment.
* Temperature >100.4°F at the time of enrollment.
* Subjects undergoing treatment for tuberculosis infection or disease.
* Having received any vaccinations or planned vaccinations with a live vaccine within 30 days prior or after study vaccination.
* Having received any vaccinations or planned vaccinations with a killed vaccine within 14 days prior or after study vaccination.
* Chronic administration of immuno-suppressant or immune-modifying drugs.
* Post organ transplant subjects whether or not receiving chronic immunosuppressive therapy.
* Administration or planned administration of immunoglobulins and/or any blood products.
* Use of any investigational or non-registered drug or vaccine.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2005-07

PRIMARY OUTCOMES:
Occurrence, relationship and intensity of any serious and/or unexpected adverse reaction at any time during the study

SECONDARY OUTCOMES:
Neutralisation assay specific seroconversion rates and geometric mean titres (at all blood sampling time points)
ELISA specific seroconversion rates and geometric mean titres (at all blood sampling time points)

CONTACTS AND LOCATIONS:
Overall Officials: Richard N Greenberg, M.D., Principal Investigator — University of Kentucky School of Medicine
Locations (5):
- United States (5):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Washington University School of Medicine, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt AIDS Clinical Trials Center, Nashville, Tennessee

REFERENCES:
- [Derived] Greenberg RN, Overton ET, Haas DW, Frank I, Goldman M, von Krempelhuber A, Virgin G, Badeker N, Vollmar J, Chaplin P. Safety, immunogenicity, and surrogate markers of clinical efficacy for modified vaccinia Ankara as a smallpox vaccine in HIV-infected subjects. J Infect Dis. 2013 Mar 1;207(5):749-58. doi: 10.1093/infdis/jis753. Epub 2012 Dec 7. PMID 23225902